CLINICAL TRIAL: NCT02481388
Title: Effect of Cardiomegaly Associated With Inspiratory Muscle Weakness on Diaphragm Thickness and Chest Wall Volume Distribution in Patients With Heart Failure
Brief Title: Optoelectronic Pletysmography and Diaphragmatic Thickness in Heart Failure Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, dbrandao, Universidade Federal de Pernambuco
Other Study IDs: jasiel02
Record Dates: First submitted 2015-06-22; First posted 2015-06-25 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Weakness Group (WG): Patients with heart failure and a maximum inspiratory pressure (MIP) <70% of predicted MIP to age, considered as inspiratory muscle weakness. Following the recruitment process, these volunteers will be evaluated by spirometry and manovacuometry. Afterwards, volunteers will be also assessed in a maximal exercise ramp test. Before and after the ramp test, the optoelectronic pletysmography will be performed to analyse the chest wall tricompartmental distribution and the shortening velocities of rib cages muscles. Also a high-definition ultrasonography will be performed to measure the right diaphragmatic cupule thickness
  Interventions: Other: Maximal exercise ramp test
- Control group (CG): Patients with heart failure and do not have a maximum inspiratory pressure (MIP) > 70% of predicted MIP to age, considered as inspiratory muscle weakness. Following the recruitment process, these volunteers will be evaluated by spirometry and manovacuometry. Afterwards, volunteers will be also assessed in a maximal exercise ramp test. Before and after the ramp test, the optoelectronic pletysmography will be performed to analyse the chest wall tricompartmental distribution and the shortening velocities of rib cages muscles. Also a high-definition ultrasonography will be performed to measure the right diaphragmatic cupule thickness
  Interventions: Other: Maximal exercise ramp test

INTERVENTIONS:
Other: Maximal exercise ramp test — The maximal exercise ramp test, symptom-limited, performed by all patients in the study was performed based on treadmill ramp protocol through ErgoPC Elite® software associated with 12-channels electrocardiogram. Respiratory variables were obtained in standard conditions of temperature, pressure and humidity (StPD), breath-by-breath, with the patient breathing through a face mask without leaks coupled to gas analyzer (Cortex - Metamax 3B, Germany).To ensure that patients reached maximum effort during the examination, only the tests which patients obtain a respiratory exchange ratio (RR) ≥1.1 were accepted .

SUMMARY:
The investigators aimed to evaluate the effects of cardiomegaly associated with inspiratory muscle weakness on tricompartmental distribution of chest wall volumes, on the thickness of the right hemidiaphragm and on the contraction speed of the respiratory muscles. As method of the present research, a pilot cross-sectional study was conducted with fourteen (14) patients with heart failure, functional class II and III, clinically stable, with cardiomegaly. Two groups were formed: one group with inspiratory muscle weakness (WG) (maximal inspiratory pressure - MIP <70% predicted MIP) and a control group without weakness (CG). The pulmonary and respiratory muscle functions were assessed by spirometry and manometer, respectively. Before and after maximal exercise test, optoelectronic plethysmography was performed to evaluate the distribution of volumes, the kinematics and the contraction speed of chest wall muscles. The high-resolution ultrasonography was also used before and after the maximum test for obtaining diaphragmatic thickness

ELIGIBILITY:
Inclusion Criteria:

* Both sexes, 18-60 years;
* Functional Class II-III according to the New York Heart Association;
* Echocardiography of the last six months showing showing left ventricular ejection fraction (LVEF) ≤ 45% measured by Teichholz method;
* Echocardiography the last six months showing cardiac hypertrophy (Diameter of Left Ventricular Diastolic (LVDD)> 54 mm, diameter of Systolic Left Ventricular (LVSD)> 34mm) 30 measured by Teichholz method;
* Optimized by the medical point of view and
* Clinical stability

Exclusion Criteria:

* Unstable angina; myocardial infarction or heart surgery up to three months before the survey;
* Orthopedic diseases, infectious or chronic metabolic diseases;
* The relation between forced expiratory volume in the first second and forced vital capacity (FEV1 / FVC) <70% of predicted characterizing obstructive respiratory disorder and
* Active smokers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic thickness | 30 minutes
  A high-definition ultrasound in the the B mode with linear transducer of 7.5 megahertz was used to measure diaphragmatic thickness. In the lateral decubitus position, the transducer was positioned perpendicular to the chest, between the eighth and ninth intercostal spaces between the right anterior and medium axillary lines. Diaphragm was identified by two hyperechoic (bright) lines parallel to the pleural and parietal membranes respectively. The measurement of diaphragm thickness was held from the middle of the pleural line to the middle of peritoneal. The average of 3 final measures taken at the apposition zone obtained: at functional residual capacity (thickness of the relaxed diaphragm - Erel) at the end of the total lung capacity (thickness of the diaphragm contracted - Econt) and during a maximal inspiratory pressure maneuver from functional residual capacity.
Chest Wall tricompartmental volumes | 30 minutes
  The images generated by the triangulation of the infra-red light reflected by 89 markers placed over volunteers' chest walls and captured by 8 cameras allows the visualization of the same thoraxes as entire structure and in its own tricompartmental division: pulmonary rib cage (RCp), abdominal rib age (RCab) and abdomen (AB). Each compartment can be evaluated in terms of their volume variation across the recorded respiratory cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Jasiel F do Nascimento Junior, Bch, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Laboratório de Fisiologia e Fisioterapia Cardiopulmonar, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Chiappa GR, Roseguini BT, Vieira PJ, Alves CN, Tavares A, Winkelmann ER, Ferlin EL, Stein R, Ribeiro JP. Inspiratory muscle training improves blood flow to resting and exercising limbs in patients with chronic heart failure. J Am Coll Cardiol. 2008 Apr 29;51(17):1663-71. doi: 10.1016/j.jacc.2007.12.045. PMID 18436118
- [Result] Brandao DC, Lage SM, Britto RR, Parreira VF, de Oliveira WA Jr, Martins SM, Aliverti A, de Andrade Carvalho L, do Nascimento Junior JF, Alcoforado L, Remigio I, de Andrade AD. Chest wall regional volume in heart failure patients during inspiratory loaded breathing. Respir Physiol Neurobiol. 2012 Mar 15;180(2-3):269-74. doi: 10.1016/j.resp.2011.12.002. Epub 2011 Dec 13. PMID 22193337
- [Result] Aliverti A, Cala SJ, Duranti R, Ferrigno G, Kenyon CM, Pedotti A, Scano G, Sliwinski P, Macklem PT, Yan S. Human respiratory muscle actions and control during exercise. J Appl Physiol (1985). 1997 Oct;83(4):1256-69. doi: 10.1152/jappl.1997.83.4.1256. PMID 9338435